CLINICAL TRIAL: NCT07046143
Title: A Study of the Efficacy of Noninvasive Spinal Cord Electrical Stimulation in Neuropathic Pain
Brief Title: Study on the Efficacy of Non-invasive Spinal Cord Electrical Stimulation in Neuropathic Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchang University Affiliated Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Wentao Zeng, Prinicipal Investigator, Nanchang University Affiliated Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFYLL-KY-PJ-2025-003
Record Dates: First submitted 2025-05-31; First posted 2025-07-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: Neuropathic Pain
Keywords: Transcutaneous spinal cord electrical stimulation; Neuropathic Pain; lumbago
MeSH Terms: conditions — Neuralgia; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): The experimental group received noninvasive spinal cord electrical stimulation treatment
  Interventions: Device: tSCS
- control group (No Intervention): The placebo control group's initial stimulation intensity was set at the sensory threshold, maintained for 30 seconds, and then gradually reduced to zero over the remaining duration.

INTERVENTIONS:
Device: tSCS — The test group received non-invasive spinal cord electrical stimulation therapy during hospitalization. Patients were positioned prone or seated, with the anode placed above the iliac crest on the affected side and the cathode covering the paravertebral region of the lumbosacral enlargement corresponding to the painful dermatome. The stimulation frequency was adjusted to 10,000 Hz, with a treatment frequency of 30 Hz and a pulse width of 1 millisecond. The waveform was square, with each treatment session lasting 20 minutes. Stimulation intensity was set to the patient's tolerable threshold. Sessions were administered twice daily, each lasting 20 minutes.
  Arms: test group

SUMMARY:
This study is a randomized, double-blind, controlled clinical trial designed to evaluate the impact of non-invasive spinal cord electrical stimulation (tSCS) on the outcome of patients with neuropathic pain.Subjects will be randomized into a test group (treated with tSCS) and a control group (receiving sham stimulation).The intervention period was during the patient's hospitalization, with a follow-up period of 3 months.Patients' pain and quality of life will be assessed at baseline, at the end of the intervention, and during the follow-up period to compare the difference in efficacy between the two groups.

DETAILED DESCRIPTION:
The study subjects were patients with low back pain caused by neuropathic pain patients, who were assessed and screened by professionally trained medical personnel according to the inclusion and exclusion criteria, and those who met the enrollment criteria signed an informed consent form after they gave their informed consent and were formally included in the study. A computerized randomization system was applied to randomly divide them into a test group and a control group.Both groups were operated with non-invasive spinal cord stimulation devices manufactured by the same company, with the test group receiving real and effective non-invasive spinal cord electrical stimulation (Device A), while the control group received placebo stimulation (Device B). Throughout the double-blind intervention, neither the subjects nor the assesseors who operated the devices were aware of the difference between the two devices (Device A and Device B) and were completely blinded.

For the subjects randomized to receive noninvasive spinal cord electrical stimulation, the unblinded researchers carried out the study according to the following research steps: ① Before the treatment, the patient's skin was wiped with 75% alcohol, and the patient was asked to take a prone or sitting position, The anode is placed above the anterior superior iliac spine on the affected side, while the cathode covers the paravertebral region of the lumbosacral enlargement corresponding to the painful dermatome.② The stimulation frequency was adjusted to 10,000Hz, the treatment frequency was 30Hz, the pulse width was 1ms, the waveform was square wave, and the duration of single treatment was 20min. ③ The test group's stimulation intensity was set at the patient's tolerable threshold. The placebo control group's initial stimulation intensity was set at the sensory threshold, maintained for 30 seconds, and then gradually reduced to zero over the remaining duration.④ The equipment was sterilized by wiping with 75% alcohol after the treatment.Subjects randomized to receive sham stimulation operated according to the above study steps, and the device output interface adjustment parameters were all consistent. Both the test group and the control group received non-invasive spinal cord electrical stimulation during hospitalization, twice daily for 20 minutes each session. During the study period, subjects in both groups received the same other conventional rehabilitation treatments.

The basic information of the patients was recorded before treatment, including gender, age, etiology, and duration of the disease.The McGill Pain Questionnaire (MPQ), Visual Analog Scale (VAS), Oswestry Dysfunction Index Questionnaire (ODI), EEG data during tSCS stimulation, Quality of Life Scale (SF-36), and Patient General ImpressionImprovement Scale (CGI-1), Pittsburgh Sleep Quality Index (PSQI), Self-Assessment Scale for Anxiety (SAS), Self-Assessment Scale for Depression (SDS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old;
* Meet the diagnostic criteria for neuropathic pain
* Chronic low back pain due to neuropathic pain, with or without leg pain;
* The skin at the site of irritation is intact;
* The patient's vital signs are stable.

Exclusion Criteria:

* Pain is mainly caused by non-neuropathic factors, such as acute inflammation and trauma;
* Those with severe mental illness affecting the study assessment, those with severe cognitive impairment unable to communicate normally or with very poor compliance;
* Accompanied by severe cardiac, hepatic, renal and other vital organ insufficiency;
* Recently received other related treatments that may affect the impact of neuropathic pain.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
McGill Pain Questionnaire | Study pre-intervention and post-intervention weeks one and two
  McGill Pain Questionnaire (MPQ): (1) The questionnaire contains two main categories, the Pain Rating Index (PRI) and the Pain Intensity (PI). (2) The PRI section consists of 20 subcategories totaling 78 descriptive words, and patients are asked to mark one word from each category that best indicates their pain (no suitable may be left unchecked), and these words indicate the different components of pain. categories 1-10 are sensory, 11-15 are affective, 16 are evaluative, and 17-20 are other.Scores are 0-78, with 0 being no pain and 78 being severe pain. (3) The PPI can be used to assess the intensity of generalized pain on a scale of 0-5, with the higher the score, the more pronounced the pain.
The Oswestry Dysfunction Index Questionnaire | Study pre-intervention and post-intervention weeks one and two
  The Oswestry Dability Index is a 10-question questionnaire consisting of 10 questions on pain intensity, self-care, lifting, walking, sitting, standing, disturbed sleep, sexuality, social life, and travel, with 6 options for each question and a maximum score of 5 for each question.The maximum score for each question is 5 points, 0 points for the first option and 5 points for the last option in that order. If all 10 questions are answered, the score is: actual score/50 (highest possible score) x 100%, and if one question is not answered, the score is: actual score/45 (highest possible score) x 100%, with higher scores indicating more severe dysfunction.
Visual Analog Scale | Study pre-intervention and post-intervention weeks one and two
  Visual analog scoring method.A 10 cm horizontal line was drawn on the paper, with 0 mm at one end of the line, indicating "no pain at all", and 10 mm at the other end, indicating "extreme pain"; the pain level increased from 0 mm to 10 mm, and the higher the score, the more intense the pain.The higher the score, the more intense the pain.
EEG | Study pre-intervention and post-intervention weeks one and two
  The recording parameters are as follows: recording bandwidth(dc-1000hz)，sampling rate (1000hz). The main measures of eeg are as follows and focued on 0.1- 40hz thus include delta, theta, alpha, beta and gamma band: qualitative waveform, power spectral density, fuctional connectivity, graph theory measurs. However, since biomarkers of pain is just one of the study objectives, we can not determine all measures that might be used in the future.

SECONDARY OUTCOMES:
Quality of Life Scale | Pre-treatment and first week, second week, 3 months, 6 months, 1 year post-treatment
  for assessing the overall quality of life of patients
Patient General Impression of Improvement Scale | Pre-treatment and first week, second week, 3 months, 6 months, 1 year post-treatment
  to assess patient self-perceived improvement in pain
Pittsburgh Sleep Quality Index | Pre-treatment and first week, second week, 3 months, 6 months, 1 year post-treatment
  assesses the quality of a patient's sleep
Self-assessment scale for anxiety | Pre-treatment and first week, second week, 3 months, 6 months, 1 year post-treatment
  assessment of the patient's psychological status. Anxiety scale: normal (<50 points); mild anxiety (50-60 points); moderate anxiety (61-70 points); severe anxiety (>70 points).
Self-assessment scale for depression | Pre-treatment and first week, second week, 3 months, 6 months, 1 year post-treatment
  Depression scale: mild depression (53-62 points); severe depression (63-72 points); severe depression (>72 points).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liang, Study Director — Affiliated Rehabilitation Hospital of Nanchang University
Locations (1):
- NanChang, Nanchang, Jiangxi, China